CLINICAL TRIAL: NCT05825222
Title: A Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy of E-PR-01 on Musculoskeletal Health in Physically Active Individuals
Brief Title: A Study to Evaluate the Efficacy of E-PR-01 on Musculoskeletal Health in Physically Active Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EB/221202/MUV/JP
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-10

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Stratified block randomization, Sequentially numbered, sealed, opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-PR-01 (Low Dose) (Active Comparator): One capsule twice a day
  Interventions: Dietary Supplement: E-PR-01 (Low dose)
- E-PR-01 (High Dose) (Active Comparator): One capsule twice a day
  Interventions: Dietary Supplement: E-PR-01 (High Dose)
- Placebo (Placebo Comparator): One capsule twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: E-PR-01 (Low dose) — One Capsule to be consumed twice a day
  Arms: E-PR-01 (Low Dose)
Dietary Supplement: E-PR-01 (High Dose) — One Capsule to be consumed twice a day
  Arms: E-PR-01 (High Dose)
Dietary Supplement: Placebo — One Capsule to be consumed twice a day
  Arms: Placebo

SUMMARY:
The present study is a randomized, placebo-controlled, parallel-group, double-blind (double-dummy) clinical study. Not more than 210 individuals will be screened, and considering a screening failure rate of 18%, approximately 168 participants will be randomized in a ratio of 1:1:1 to receive E-PR-01 (LD: 200 mg/day), E-PR-01 (HD: 400 mg/day), or placebo (400 mg/day). After accounting for a dropout/withdrawal rate of 15%, each group will have at least 48 completed participants with equal numbers of participants having knee and lumbo-sacral as index joint. The intervention duration for all the study participants will be approximately 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Males & females aged 40-60 years with history of knee and/or low back pain aggravation on physical stress (squatting, walking, running, and cycling) for at least 3 months and maximum up to 3 years.
* BMI ≥24.9 to ≤29.9 kg/m2.
* Participants with either of the following two criteria:

  1. On screening, low back pain score ≥60 on a 100-point P-NRS after completion of 4 sets of five-repetition sit-to-stand test along with radiological evidences of lumbo-sacral degeneration indicated by 2 or more of the following:

     i. Loss of lordosis ii. Joint space narrowing iii. Presence of osteophytes iv. Bony spurs
  2. On screening, knee joint pain score ≥60 on a 100-point P-NRS after completion of 4 sets of five-repetition sit-to-stand test along with radiological evidences of knee degeneration indicated by doubtful narrowing of the joint space, possible osteophytes, or definite small osteophytes, definite narrowing of the joint space.
* Participants with a score of ≤30 on the MSK-HQ scale.
* Moderate physical activity level as assessed by International Physical Activity Questionnaire (IPAQ)-Short form.
* Willingness to participate in the study and comply with the study procedures and required visits.
* Has the ability to understand and sign a written informed consent form, which must be completed prior to study specific tasks being performed.
* Must be literate and have the ability to complete the study-based questionnaires and tasks.
* Ready to refrain from intake of analgesics one week prior to screening visit and during the study.
* Female participants of childbearing age must be willing to use the accepted methods of contraception during the study.

Exclusion Criteria:

* P-NRS score >40 points on rest.
* Any other type of pain except joint pain including muscular, nervine or pain due to acute injury.
* For knee joint, participants with the radiographic evidence of no presence of OA, or multiple moderately sized osteophytes with definite JSN, sclerosis, or definite bony deformity will be excluded.
* For lumbo-sacral joint, participants with the radiographic evidence of normal, or disc space narrowing with osteophytes, or bone sclerosis, disc space narrowing, large osteophytes will be excluded.
* Known cases of osteoporosis.
* Current intake of disease modifying antirheumatic drugs for joint pain.
* Participants with neurological characteristic of pain (shooting, burning, stabbing, or electric shock-like pain, tingling, numbness, or a "pins and needles" feeling).
* Participants suffering from insomnia and restless leg syndrome.
* Participants with uncontrolled hypertension (defined as systolic blood pressure (SBP)≥140 mm Hg and/or diastolic blood pressure (DBP) ≥90 mm Hg despite anti-hypertensive treatment).
* Participants suffering from uncontrolled type II diabetes mellitus (Random blood glucose (RBG)≥200 mg/dl (11.1 mmol/l) despite anti-diabetic treatment).
* History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders.
* History of hyperacidity with at least one episode/week.
* History of use of any dietary supplement within 2 weeks of screening visit.
* Heavy drinkers defined as - for men, consuming more than 4 drinks on any day or more than 14 drinks per week and for women, consuming more than 3 drinks on any day or more than 7 drinks per weekly.
* Participants who have any other diagnosed disease or condition, or are using any medication, that in the judgment of the investigator would puthim/ her at unacceptable risk for participation in the study or may interfere with evaluations in the study or noncompliance with intervention or visits.
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
* Participants who have had participated in a study of an investigational product 90 days prior to the screening.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of E-PR-01 (Low Dose and High Dose) on the musculoskeletal health as assessed by the Musculoskeletal Health Questionnaire (MSK-HQ) compared to baseline and placebo. | Day 90
  The MSK-HQ is a short 14 item questionnaire that allows people with musculoskeletal conditions to report their symptoms and quality of life. The total score ranges from 0-56, with 56 being the best possible musculoskeletal health state.
To evaluate the effect of E-PR-01 (Low Dose and High Dose) on the musculoskeletal health as assessed by the Musculoskeletal Health Questionnaire (MSK-HQ) compared to baseline and placebo. | Day 60
  The MSK-HQ is a short 14 item questionnaire that allows people with musculoskeletal conditions to report their symptoms and quality of life. The total score ranges from 0-56, with 56 being the best possible musculoskeletal health state.
To evaluate the effect of E-PR-01 (Low Dose and High Dose) on the musculoskeletal health as assessed by the Musculoskeletal Health Questionnaire (MSK-HQ) compared to baseline and placebo. | Day 30
  The MSK-HQ is a short 14 item questionnaire that allows people with musculoskeletal conditions to report their symptoms and quality of life. The total score ranges from 0-56, with 56 being the best possible musculoskeletal health state.

SECONDARY OUTCOMES:
To evaluate the effect of 90 days' administration of E-PR-01 (LD and HD) on Pain Numeric Rating Scale (P-NRS) compared to baseline and placebo. | Day 7, 30, and 90
  Pain numeric rating scale (P-NRS) score is taken after 4 sets of five-repetition sit-to-stand test. It is a unidimensional measure of pain intensity in adults. It is a single 11-point numeric scale with 0 indicating one pain extreme (eg: "no pain") and 100 indicating the other pain extreme (eg: "worst pain imaginable").
To evaluate the effect of 90 days' administration of E-PR-01 (LD and HD) on Range of motion (ROM) of the index joint compared to baseline and placebo. | Day 90
  This assessment will be done with the use of a manual Goniometer and the angle will be measured in degrees.
To evaluate the effect of 90 days' administration of E-PR-01 (LD and HD) on Quality of life (QoL) compared to baseline and placebo. | Day 30 and 90
  This is assessed by the change in Euro QoL 5 dimension 5 level (EQ-5D-5L) questionnaire score. The EQ VAS records the respondent's self-rated health on a vertical VAS numbered from 0-100 where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
To evaluate the effect of 90 days' administration of E-PR-01 (LD and HD) on Rescue Medication consumption. | Day 30 and 90
  Proportion of participants who used rescue medication (RM) during the study compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shalini Srivastava, MBBS, MD, Principal Investigator — Vedic Lifesciences Pvt. Ltd.
Locations (6):
- India (6):
  - Proactive Orthopedic Clinic, Mumbai, Maharashtra
  - Ayush Nursing Home, Mumbai, Maharashtra
  - Diamond Orthopedic Multispeciality Hospital, Mumbai, Maharashtra
  - Sankalp Ortho Clinic, Nashik, Maharashtra
  - O2 Clinic Orthopaedics and Opthalmology, Nashik, Maharashtra
  - Sparsh Hospital, Panvel, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided